CLINICAL TRIAL: NCT03295136
Title: Impact of Health Promotion Course for Female Employees on Health Promotion in the Work Place.
Brief Title: Impact of Employee Health Promotion Course on Health Promotion in the Work Place.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRK-HMO-CTIL
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Lifestyle Risk Reduction; Health Knowledge, Attitudes, Practice; Empowerment
MeSH Terms: conditions — Risk Reduction Behavior; Behavior; Empowerment

STUDY DESIGN:
Intervention Model Description: This study includes a pre/post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Promotion Training for Women Employees (Experimental): Groups of women employees will participate in a 20 session health promotion training course. The course will include health education and health promotion knowledge and skills, as well as leadership and project building skills, including empowerment, change process, recruiting partners and more. The first 15 sessions will be weekly session, while the remaining five will take place every couple of months throughout the following year.
  Interventions: Behavioral: Health Promotion Training for Women Employees

INTERVENTIONS:
Behavioral: Health Promotion Training for Women Employees — Group intervention over a one year, acquiring health promotion tools and skills, as well as leadership and project designing and implementation skills.

SUMMARY:
People of working age spend most of their day at work, and usually have less time to participate in other activities, the work day in Israel being one of the longest in the OECD. Work places, therefore, present the most suitable setting for health interventions, as they are an accessible and available framework and have real potential of creating change.

The current Health Promotion in the Work Place training course aims to train female employees to design, implement, and evaluate a health promotion program in their workplace, as well as promote personal change in improving healthy habits, and empowering the participants. A unique course has been designed, consisting of 20 sessions- 15 consecutive sessions, and 5 maintenance sessions throughout the year. The course will focus on acquiring health knowledge and health promotion skills, as well as leadership skills and empowerment.

DETAILED DESCRIPTION:
Poor health of employees can cause absences, lack of continuous service, decreased output or productions, fatigue or lack of concentration, and eventually financial damage to the employer. Research shows that health promotion programs in the work place improve employee's physical and emotional health, as well as their sense of commitment, belonging, and responsibility.

People of working age spend most of their day at work, and usually have less time to participate in other activities, the work day in Israel being one of the longest in the OECD. Work places, therefore, present the most suitable setting for health interventions, as they are an accessible and available framework and have real potential of creating change.

The current Health Promotion in the Work Place training course aims to train female employees to design, implement, and evaluate a health promotion program in their workplace, as well as promote personal change in improving healthy habits, and empowering the participants. Objectives include improving eating habits, increasing engagement in physical activity, increasing self-efficacy, and designing a detailed health promotion program in the work place, based on it's needs, and implementing it there.

In order to accomplish these objectives, a unique course has been designed, consisting of 20 sessions- 15 consecutive sessions, and 5 maintenance sessions throughout the year. The course will focus on acquiring health knowledge and health promotion skills, as well as leadership skills and empowerment. The participants will learn how to build programs, market them to their coworkers and employers, budget them, recruit partners, create a Gantt charts, implement and evaluate. The maintenance sessions will take place in different work places, so that the participants can showcase their projects.

Data will be collected at baseline and 2 post interventions follow up points (after 15 weeks and after one year).

ELIGIBILITY:
Inclusion Criteria:

* Female employees from governmental offices and private organizations, willingness to commit to participation in the health promotion training course and lead a health promotion project in their place of work, willingness to make make personal change.

Exclusion Criteria:

* None.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in Nutrition Habits | At baseline, 15 weeks after intervention initiation, and one year post intervention.
  Participants complete self report survey indicating their eating habits, including consumption of sweets, sweet beverages, fruits and vegetables, whole grains, and legumes.
Change in Physical Activity Habits | At baseline, 15 weeks after intervention initiation, and one year post intervention.
  Participants complete self report survey indicating their physical activity habits, including minutes of engaging in vigorous and moderate physical activity. Measures will include average daily minutes of engaging in physical activity, and adherence to WHO recommendation (150 minutes of moderate physical activity a week, or 75 minutes of vigorous physical activity a week).
Health Promotion projects in the Work Place | One year post intervention
  Each participant will have implemented a health promotion project in their workplace, according to the timeline and goals defined in each project. This will be assessed through phone interviews with the participants.

SECONDARY OUTCOMES:
Change in Self Efficacy | At baseline, 15 weeks after intervention initiation, and one year post intervention.
  Self Efficacy will be assessed through self report questionnaires, assessing participants self efficacy regarding their leadership skills, ability to implement a health promotion project, create partnerships, evaluate a project, and influence women in their community.
Change in cardiovascular disease knowledge | At baseline, 15 weeks after intervention initiation, and one year post intervention.
  Cardiovascular disease knowledge will be assessed through a self report questionnaire based on the American Heart Association's Cardiovascular disease knowledge survey items

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Isreal, Jerusalem, Israel

REFERENCES:
- [Background] Baxter S, Sanderson K, Venn AJ, Blizzard CL, Palmer AJ. The relationship between return on investment and quality of study methodology in workplace health promotion programs. Am J Health Promot. 2014 Jul-Aug;28(6):347-63. doi: 10.4278/ajhp.130731-LIT-395. PMID 24977496
- [Background] VanWormer JJ, Boucher JL, Sidebottom AC. Two-year impact of lifestyle changes on workplace productivity loss in the Heart of New Ulm Project. Occup Environ Med. 2015 Jun;72(6):460-2. doi: 10.1136/oemed-2014-102620. Epub 2015 Apr 9. PMID 25858035
- [Background] Leigh JP. Economic burden of occupational injury and illness in the United States. Milbank Q. 2011 Dec;89(4):728-72. doi: 10.1111/j.1468-0009.2011.00648.x. PMID 22188353
- [Derived] Greenberg KL, Donchin M, Leiter E, Zwas DR. Health ambassadors in the workplace: a health promotion intervention mobilizing middle managers and RE-AIM evaluation of outcomes. BMC Public Health. 2021 Aug 23;21(1):1585. doi: 10.1186/s12889-021-11609-8. PMID 34425815